CLINICAL TRIAL: NCT06902961
Title: The Effects of Game-Based Exercises on Balance, Kinesiophobia, Fatigue Levels, and Pain in Sedentary Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-01/06
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Sedentary Behavior
Keywords: pain; exercise
MeSH Terms: conditions — Sedentary Behavior; Pain; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game-based exercise group (Experimental): game-based
  Interventions: Other: Game-based exercise group
- control group (Active Comparator): control group
  Interventions: Other: control group

INTERVENTIONS:
Other: Game-based exercise group — Game-based exercise group
  Arms: Game-based exercise group
Other: control group — control group
  Arms: control group

SUMMARY:
Physical activity is a significant factor that greatly affects human health. However, with the development of technology, there has been a significant decrease in the physical activity levels of individuals in their daily lives, leading to the emergence of a sedentary society.

DETAILED DESCRIPTION:
Technological advancements, such as electronic devices and machines that replace human labor, push individuals toward laziness, encouraging them to adopt a more inactive lifestyle.

ELIGIBILITY:
Inclusion Criteria

* Accepting to participate in the study
* Between the ages of 18 and 45
* Physical activity level according to the International Physical Activity Questionnaire (short form) between 600 MET- 1500 MET min/week
* Having an appropriate cognitive level (not having a cognitive level that would make it difficult to understand the study or to perform the exercise) Exclusion Criteria
* Physical activity level >1500 MET-min/week according to the International Physical Activity Questionnaire (short form)
* Having cancer and malignant tumours
* Presence of cognitive problems
* Severe vision problems (colour blindness, blindness, etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Single Leg Stance Test | 6 weeks
  A method used to assess static balance. Participants are asked to stand on one leg with eyes open and arms crossed at chest level. The raised leg should not touch or make contact with the ground. The individual must maintain their position without any jerking, jumping, or touching any nearby objects for support. The time they can maintain the position is recorded in seconds.
Libra Swivel Balance Board | 6 weeks
  A computer-based device used to assess dynamic balance. The Libra swivel balance board (42 cm long and 42 cm wide) is equipped with a computer system. Dynamic balance is measured using specific software
International Physical Activity Questionnaire | 6 weeks
  this questionnaire provides information on the time spent on sitting, walking, moderate-intensity, and vigorous-intensity activities. The Turkish validity and reliability study was conducted by Öztürk (2005). It classifies individuals as sedentary, minimally active, or highly active based on MET-minute/week score
Tampa Kinesiophobia Scale | 6 weeks
  It evaluates fear of movement and injury. The scale consists of 17 items with 4 response options (1 = Strongly Disagree to 4 = Strongly Agree). Higher scores indicate greater kinesiophobia
Fatigue Severity Scale | 6 weeks
  This scale measures the severity of fatigue over the last week, with 9 questions scored on a 7-point scale. Higher scores (28 or above) indicate severe fatigue.
McGill Pain Questionnaire | 6 weeks
  Developed by Melzack, this scale assesses pain sensory aspects using 15 descriptive words. Participants rate their pain intensity on a scale from 0 (none) to 3 (severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Bahceşehir University Health Center, Istanbul, Turkey (Türkiye)